CLINICAL TRIAL: NCT02729961
Title: A Phase I/II Open-Label Dose-Finding Study of Ceritinib Combined With Brentuximab Vedotin for Front-Line Treatment of ALK-Positive Anaplastic Large Cell Lymphoma
Brief Title: Ceritinib With Brentuximab Vedotin in Treating Patients With ALK-Positive Anaplastic Large Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administrative closure
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9522; NCI-2016-00396 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9522 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive; CD30-Positive Neoplastic Cells Present; Systemic Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — Brentuximab Vedotin; ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (brentuximab vedotin, ceritinib) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1. Patients also receive ceritinib PO QD on days 8-21 of course 1 and on days 1-21 for all subsequent courses. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Ceritinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Ceritinib — Given PO
  Other Names: LDK 378; LDK378; Zykadia
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of ceritinib when given together with brentuximab vedotin to see how well they work in treating treatment-naive patients with anaplastic lymphoma kinase (ALK)-positive anaplastic large cell lymphoma. Ceritinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as brentuximab vedotin, may interfere with the ability of tumor cells to grow and spread. Giving ceritinib together with brentuximab vedotin may be a better treatment for ALK-positive anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To define a dose of ceritinib administered concurrently with brentuximab vedotin that has an acceptable toxicity profile (based on dose-limiting toxicity [DLT] rate) and sufficient efficacy (based on response rate) among patients with treatment-naive ALK-positive anaplastic large cell lymphoma (ALCL). SECONDARY OBJECTIVES: I. To assess the antitumor activity of ceritinib and brentuximab vedotin combination in treatment-naive patients with ALK-positive ALCL. II. To assess the utility of the molecular marker of ALK-positive ALCL in patient's plasma before, during and after therapy for disease risk assessment and post-treatment monitoring. OUTLINE: This is a phase I, dose-escalation study of ceritinib followed by a phase II study. Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1. Patients also receive ceritinib orally (PO) once daily (QD) on days 8-21 of course 1 and on days 1-21 for all subsequent courses. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 3 months up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive systemic ALK-positive ALCL patients
* Histologically confirmed diagnosis of cluster of differentiation (CD)30-positive ALCL with documented ALK-positive status
* Fluorodeoxyglucose (FDG)-avid disease by positron emission tomography (PET) and dimensional measurable disease of at least 1.5 cm as documented by radiographic technique (spiral computed tomography [CT] preferred)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Absolute neutrophil count (ANC) >= 1500/ul
* Platelet count >= 75,000/ul (unless documented bone marrow involvement with lymphoma)
* Hemoglobin (Hgb) >= 8 gr/dL
* Serum creatinine =< 1.5 x mg/dL and/or calculated creatinine clearance (using Cockcroft-Gault formula) >= 30 mL/min
* Total bilirubin =< 1.5 x upper limit of normal (ULN), except for patients with Gilbert's syndrome or documented hepatic involvement with lymphoma who may be included if bilirubin =< 3.0 x ULN or direct bilirubin =< 1.5 x ULN
* Aspartate transaminase (AST) =< 3 x ULN, except with liver involvement by the lymphoma who are only included if AST =< 5 x ULN; alanine transaminase (ALT) < 3.0 x ULN, except with liver involvement by the lymphoma who are only included if AST =< 5 x ULN
* Alkaline phosphatase (ALP) =< 5.0 x ULN
* Fasting plasma glucose =< 175 mg/dL (=< 9.8 mmol/L)
* Serum amylase =< 2 x ULN
* Serum lipase =< ULN
* Patients must have the following laboratory values or have the following laboratory values corrected to be within normal limits before the first dose of ceritinib: * Potassium * Magnesium * Phosphorus * Total calcium (corrected for serum albumin)
* Females of child bearing potential, defined as all women physiologically capable of becoming pregnant, must have a negative serum or urine beta human chorionic gonadotropin (b-hCG) pregnancy test results within 7 days prior to the first dose of study treatment, and must agree to use highly effective methods of contraception during dosing and for 3 months after the last dose of study treatment; highly effective methods of contraception include: * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment * Male sterilization (at least six months prior to screening) with the appropriate post-vasectomy documentation of absence of sperm in the ejaculate; for female subjects on the study the vasectomized male partner should be sole partner for that subject * Combination of any two of the following: ** Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception ** Placement of an intrauterine device (IUD) or intrauterine system (IUS) ** Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository * In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or who have had a bilateral tubal ligation or hysterectomy
* Sexually active males must agree to use a condom during intercourse while receiving and for 3 months after the last dose of study treatment; male patients should not father a child for 3 months after the last dose of study treatment; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
* Patients or their legally authorized representative must have the ability to understand and provide signed informed written consent
* Patients must express willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures

Exclusion Criteria:

* Known hypersensitivity to any of the excipients of ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate)
* Known prior history of interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention)
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of ceritinib (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome) or inability to swallow up to five ceritinib capsules daily
* History of pancreatitis or history of increased amylase or lipase that was due to pancreatitis
* Other severe, acute, or chronic medical condition including uncontrolled diabetes mellitus or psychiatric condition or laboratory abnormalities that, in the opinion of the investigator, may increase risk associated with study participation or may interfere with the interpretation of study results
* Major surgery (e.g. intra-abdominal, intra-thoracic or intra-pelvic) within 4 weeks prior to starting study treatment or lack of recovery from side effects of such procedure; video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can receive study treatment >= 1 week after these procedures
* History of another primary malignancy that has not been in remission for at least 3 years (the following malignancies are exempt from the 3 year limit: non-melanoma skin cancer, fully-excised melanoma in situ [stage 0], curatively treated, localized prostate cancer, and cervical carcinoma in situ in biopsy or a squamous intraepithelial lesion on Papanicolau [PAP] smear)
* Known cerebral/meningeal disease
* Clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as: * Unstable angina * Myocardial infarction * History of documented congestive heart failure (New York Heart Association functional classification III-IV) * Uncontrolled hypertension defined by a systolic blood pressure (SBP) >= 160 mm Hg and/or diastolic blood pressure (DBP) >= 100 mm Hg, with or without antihypertensive medication * Ventricular arrhythmias, or supraventricular/nodal arrhythmias not controlled with medications; other cardiac arrhythmias not controlled with medications * Left ventricular ejection fraction < 20% corrected QT (QTcF) > 470 ms using Fridericia's correction on the screening electrocardiogram (ECG) * Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
* Any active grade 3 or higher (per the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 4.03) viral, bacterial, or fungal) infection within two weeks prior to the first dose of study treatment
* Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with ceritinib and for the duration of participation: * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes * Strong inhibitors or strong inducers of cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, and/or cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9) * Therapeutic doses of warfarin sodium (Coumadin) or any other Coumadin-derived anti-coagulant; anticoagulants not derived from warfarin are allowed (e.g., dabigatran, rivaroxaban, apixaban) * Unstable or increasing doses of corticosteroids; if patients are on corticosteroids for endocrine deficiencies or tumor-associated symptoms (non-central nervous system [CNS]), dose must have been stabilized (or decreasing) for at least 5 days before first dose of study treatment * Enzyme-inducing anticonvulsive agents * Herbal supplements
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive b-hCG laboratory test

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate defined as the proportion of patients with CR according to the revised Response Criteria for Malignant Lymphoma | Up to 3 years
Maximum tolerated dose (MTD) of ceritinib and brentuximab vedotin based on incidence of dose limiting toxicity (DLT) assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 6 weeks
Objective response rate defined as the proportion of patients with complete response (CR) or partial response (PR) according to the revised Response Criteria for Malignant Lymphoma | Up to 3 years
  Assessed using clinical assessment and computed tomography (CT)/positron emission tomography (PET) scans.

SECONDARY OUTCOMES:
Incidence of adverse events as assessed by NCI CTCAE version 4.03 | Up to 30 days
Laboratory abnormalities as assessed by NCI CTCAE version 4.03 | Up to 3 years
Overall survival (OS) | From start of study treatment to date of death due to any cause, assessed up to 3 years
Progression-free survival (PFS) | From start of treatment to first documentation of objective tumor progression or to death due to any cause, whichever comes first, assessed up to 3 years
  Evaluate tumor lesion size in the determination of PFS by using Revised Response Criteria for Malignant Lymphoma (modified Cheson, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Shustov, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No